CLINICAL TRIAL: NCT02530996
Title: Systemic Sclerosis (SSc) Vasculopathy: Improved Clinical Monitoring and Treatment
Acronym: Scleroderma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IMMA-006-14F
Record Dates: First submitted 2015-07-29; First posted 2015-08-21 (Estimated); Results first posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Rheumatologic Disease
MeSH Terms: conditions — Collagen Diseases | interventions — sapropterin

STUDY DESIGN:
Intervention Model Description: Twelve systemic sclerosis SSc patients were studied 5 hours after oral BH4 administration (10 mg/kg body weight) or placebo on separate days using controlled, counterbalanced, double-blind, crossover experimental design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Drug was dispensed by the investigational drug services. A controlled, counter-balanced, double-blind, crossover experimental design with two conditions, BH4 and placebo, was employed. There was a washout period of at least 5 days before crossing over into the alternate condition. On
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo before BH4 (Experimental): Six SSc received oral placebo 10 mg/kg and had flow mediated dilatation measured. After a five day washout they crossed over to oral BH4 10 mg/kg and had flow mediated dilatation measured. Blood samples were obtained from these SSc patients and assessed for oxidative stress.
  Interventions: Drug: BH4; Diagnostic Test: Vasculopathy assessment; Drug: Placebo
- BH4 before Placebo (Experimental): Six SSc received oral BH4 10 mg/kg and had flow mediated dilatation measured. After a five day washout they crossed over to oral placebo 10 mg/kg and had flow mediated dilatation measured. Blood samples were obtained from these SSc patients and assessed for oxidative stress.
  Interventions: Drug: BH4; Diagnostic Test: Vasculopathy assessment; Drug: Placebo

INTERVENTIONS:
Drug: BH4 — BH4 10 mg/kg/day given once to a total of 12 SSc patients
  Other Names: Kuvan
Diagnostic Test: Vasculopathy assessment — Non-invasive technique, flow mediated dilatation (FMD) to define vasculopathy in SSc.
  Other Names: Kuvan
Drug: Placebo — On the experimental days, patients reported to the laboratory after having consumed a standardized breakfast and oral BH4 (10mg/kg) or placebo five hours prior to their arrival. All measurements were taken at the same time of day to eliminate any diurnal effects. All participants abstained from alcohol, caffeine, and exercise for ≥12 hours prior to the study. Additionally, vasodilatory medications were discontinued 12 hours prior to study visit. In premenopausal women, measurements were performed during the early follicular phase of the menstrual cycle. All measurements were made under quiet, comfortable, ambient (~22°C) laboratory conditions.
  Other Names: Placebo from IDS

SUMMARY:
Systemic sclerosis (SSc; scleroderma) is a multi-organ systemic disease characterized by activation of immune cells, which results in vascular dysfunction (vasculopathy) and subsequent scarring (fibrosis). SSc has a higher than expect prevalence in the US military. On a national level there are 5,766 SSc patients (ICD-9 710.1) presently cared for in the Veterans Health Administration (VHA). While there is no cure for SSc, studies of therapeutics that can help slow disease progression are valuable to our Veterans. This proposal addresses the solicitation for projects with attention to SSc requested by President Obama after reviewing potential contamination of water at Camp Lejeune. This proposal is a patient-centered outreach for our Veterans with SSc to inform and prevent catastrophic endstage vascular abnormalities, including digital ulcers, pulmonary arterial hypertension (PAH) and scleroderma renal crisis in SSc. The study proposes a novel application of a therapeutic for this disease. A better understanding of the initiating insult and natural progression of SSc vasculopathy is needed in order to develop therapeutics with a goal of curing/treating the underlying disease. This project has the potential to impact not only Veterans with SSc, but also those with vascular abnormalities including digital ulcers, PAH, and renal crisis. This proposal represents a potential major therapeutic advance for our Veterans with SSc.

DETAILED DESCRIPTION:
Although SSc is heterogeneous in the extent of organ involvement and prognosis, it is accepted that all SSc cases have a progressive and usually devastating course. Since vasculopathy precedes fibrosis in this disease, a focus on understanding its natural history and preventative measures for vascular dysfunction has profound implications. This pilot work suggests that measurement of endothelial dysfunction with flow mediated dilatation (FMD) holds promise as novel method to assess disease progression as well as the therapeutic efficacy of the pharmacologic compound tetrahydrobiopterin (BH4) in SSc. The investigators believe that BH4, which targets the endothelium, has great promise to reduce SSc-related tissue hypoxia, end organ damage, and potentially may impact underlying disease progression. The first aim will adopt an integrative approach and validate a novel, non-invasive technique, FMD to define vasculopathy in SSc. The second aim and third aim (which is reported in this PRS report) will examine if BH4 is effective in ameliorating vascular dysfunction in patients with SSc and determine the role of oxidative stress in BH4-mediated improvements in vascular function in patients with SSc. The overarching goal of these aims is to improve vasculopathy detection and management in Veterans with SSc.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic sclerosis (SSc, scleroderma) by ACR/EULAR 2013 criteria.

Exclusion Criteria:

* Age < 18
* Pregnant or breast feeding
* Unwillingness to consent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy M. Frech, MD MS, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 156 patients were enrolled and screened in IRB 38705 during the funding period 01/01/2016 - 12/31/2020 in SSc clinic, but only 12 participated in a controlled, counter-balanced, double-blind, crossover experimental design with two conditions, BH4 and placebo IRB 40212 in the Utah Vascular Research Laboratory at the Salt Lake VAMC.
Pre-assignment Details: While 32 participants were intended, this study was concluded after 12 participants due to budgetary restrictions.
Groups:
- 6 SSc Patients Received BH4 Then Placebo; 6 SSc Patients Received Placebo Then BH4: Prior to January 18, 2017, a controlled, counter-balanced, double-blind, crossover experimental design with two conditions, BH4 and placebo, was employed. There was a washout period of at least 5 days before crossing over into the alternate condition.
Period: First Intervention
Arm/Group | 6 SSc Patients Received BH4 Then Placebo | 6 SSc Patients Received Placebo Then BH4
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout (5 Days)
Arm/Group | 6 SSc Patients Received BH4 Then Placebo | 6 SSc Patients Received Placebo Then BH4
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | 6 SSc Patients Received BH4 Then Placebo | 6 SSc Patients Received Placebo Then BH4
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 12 SSc Patients Received BH4 and Placebo: 12 SSc received BH4 intervention (blinded) and placebo in a cross-over design.
  Patients were studied 5 hours after oral BH4 administration (10 mg/kg body mass) or placebo on separate days using controlled, counterbalanced, double-blind, crossover experimental design
  Vasculopathy assessment: Non-invasive technique, flow mediated dilatation (FMD) to define vasculopathy in SSc.
Arm/Group | 12 SSc Patients Received BH4 and Placebo
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [59 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Dilatation (FMD)-Diameter of Artery
Description: FMD diameter of artery (mm, higher better)
Time Frame: FMD was obtained on a single day at two different time points (after placebo and intervention) after a 5 day washout period.
Measure: Mean (Standard Error); unit: mm
Groups:
- 12 SSc Participants With Placebo; 12 Participants With BH4: 12 patients were studied 5 hours after oral BH4 administration (10 mg/kg body mass) or placebo on separate days using controlled, counterbalanced, double-blind, crossover experimental design.
Arm/Group | 12 SSc Participants With Placebo | 12 Participants With BH4
Number analyzed (Participants) | 12 | 12
mm | 3.79 (0.20) | 3.78 (0.21)

2. Primary Outcome: Flow Mediated Dilatation-shear Rate
Time Frame: FMD was obtained on a single day at two different time points (after placebo and intervention) after a 5 day wash out period.
Population: Twelve patients with SSc had FMD parameters quantified after cuff at baseline, after placebo, and after BH4. FMD is expressed as a percent increase in diameter from baseline.
Measure: Mean (Standard Error); unit: sec^-1
Groups:
- 12 SSc Participants After Placebo; 12 SSc Participants After BH4: Twelve SSc patients were studied 5 hours after oral BH4 administration (10 mg/kg body mass) or placebo on separate days using controlled, counterbalanced, double-blind, crossover experimental design.
Arm/Group | 12 SSc Participants After Placebo | 12 SSc Participants After BH4
Number analyzed (Participants) | 12 | 12
sec^-1 | 95 (12) | 100 (13)
Statistical Analysis 1: Comparison: 12 SSc Participants After Placebo vs 12 SSc Participants After BH4; Statistics were performed using SPSS software (IBM, Chicago, IL). Paired t-tests were used to identify significant changes in measured variables between placebo and BH4. Unpaired t-tests were used to identify significant changes in measured variables between ordered groups. Based on data published in PMID: 25511849 power calculations for this study of SSc patients were made; Test type: Other — Power calculations were performed using G*Power computer software version 3. Sample-size calculations were based on the number of patients needed to detect significant differences in FMD between placebo and BH4; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 1.5

3. Primary Outcome: Flow Mediated Dilatation- Blood Velocity
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | 12 SSc Participants After Placebo | 12 SSc Participants After BH4
Number analyzed (Participants) | 12 | 12
cm/sec | 4.4 (0.6) | 4.5 (0.4)

4. Primary Outcome: Flow Mediated Dilatation-blood Flow
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: ml/min
Arm/Group | 12 SSc Participants After Placebo | 12 SSc Participants After BH4
Number analyzed (Participants) | 12 | 12
ml/min | 32 (7) | 30 (3)

5. Secondary Outcome: Oxidative Stress Measurement-MDA: Malondialdehyde
Description: MDA (lower better). Plasma malondialdehyde assessed by Oxis Research/Percipio Bioscience, Foster City, CA.
Time Frame: Oxidative stress measurements were obtained on a single day at two different time points (after placebo and intervention) after a 5-day wash out period.
Measure: Mean (Standard Error); unit: uM
Groups:
- 12 SSc Patients Oxidative Stress After Placebo; 12 SSc Patients Oxidative Stress After BH4: Blood samples were obtained from the antecubital patients with SSc. Serum and plasma samples were stored at -80°C until analysis. Oxidative stress was assessed by quantifying plasma malondialdehyde (MDA) (Oxis Research/Percipio Bioscience, Foster City, CA) and protein carbonyl levels (Northwest Life Science Specialties, LLC Vancouver, WA). Endogenous antioxidant capacity, assessed by superoxide dismutase (SOD) and catalase (CAT) activity, were assayed in the plasma (Cayman Chemical Company, Ann Arbor, MI). Additionally, total antioxidant capacity was assessed by measuring the ferric reducing ability of plasma (FRAP), using the method described by Benzie and Strain (17). Systemic inflammation was assessed by determining IL-6, TNF-α (18) and C-reactive protein (CRP) in serum (R&D Systems, Minneapolis, MN).
Arm/Group | 12 SSc Patients Oxidative Stress After Placebo | 12 SSc Patients Oxidative Stress After BH4
Number analyzed (Participants) | 12 | 12
uM | 2.8 (0.1) | 2.9 (0.2)

6. Secondary Outcome: Oxidative Stress Measurement-catalase (CAT)
Description: CAT (higher better) assessed by Cayman Chemical Company, Ann Arbor, MI.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: nM/min/mL
Arm/Group | 12 SSc Patients Oxidative Stress After Placebo | 12 SSc Patients Oxidative Stress After BH4
Number analyzed (Participants) | 12 | 12
nM/min/mL | 86 (7) | 78 (11)

7. Secondary Outcome: Oxidative Stress Measurement- Protein Carbonyl
Description: Protein carbonyl (lower better). Plasma protein carbonyl levels assessed by Northwest Life Science Specialties, LLC Vancouver, WA.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: nM/mg
Arm/Group | 12 SSc Patients Oxidative Stress After Placebo | 12 SSc Patients Oxidative Stress After BH4
Number analyzed (Participants) | 12 | 12
nM/mg | 0.17 (0.01) | 0.16 (0.01)

8. Secondary Outcome: Oxidative Stress Measurement- Ferric Reducing Ability of Plasma (FRAP)
Description: FRAP (higher better). FRAP assessed using the method described by Benzie and Strain.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: nM/L
Arm/Group | 12 SSc Patients Oxidative Stress After Placebo | 12 SSc Patients Oxidative Stress After BH4
Number analyzed (Participants) | 12 | 12
nM/L | 1.8 (0.1) | 1.8 (0.2)

9. Secondary Outcome: Oxidative Stress Measurement- Superoxide Dismutase (SOD)
Description: SOD (higher better). SOD assessed by Cayman Chemical Company, Ann Arbor, MI.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: U/mL
Arm/Group | 12 SSc Patients Oxidative Stress After Placebo | 12 SSc Patients Oxidative Stress After BH4
Number analyzed (Participants) | 12 | 12
U/mL | 10.7 (0.6) | 11.1 (1.3)

10. Secondary Outcome: Oxidative Stress Measurement- Interleukin 6 (IL-6)
Description: IL-6 (lower better), assessed by R&D Systems, Minneapolis, MN.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | 12 SSc Patients Oxidative Stress After Placebo | 12 SSc Patients Oxidative Stress After BH4
Number analyzed (Participants) | 12 | 12
pg/mL | 1.3 (0.5) | 1.4 (0.5)

11. Secondary Outcome: Oxidative Stress Measurement- Tumor Necrosis Factor Alpha (TNF-α,
Description: TNF-α (lower better), assessed by R&D Systems, Minneapolis, MN.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | 12 SSc Patients Oxidative Stress After Placebo | 12 SSc Patients Oxidative Stress After BH4
Number analyzed (Participants) | 12 | 12
pg/mL | 1.1 (0.2) | 1.3 (0.2)

12. Secondary Outcome: Oxidative Stress Measurement- C-reactive Protein (CRP)
Description: CRP (lower better). CRP assessed by R&D Systems, Minneapolis, MN.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | 12 SSc Patients Oxidative Stress After Placebo | 12 SSc Patients Oxidative Stress After BH4
Number analyzed (Participants) | 12 | 12
mg/L | 3.2 (0.7) | 3.1 (0.6)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 6 month for 12 patients that received BH4 and placebo.
Description: Patients were assessed on day of intervention and at their follow-up care visits for any untoward or unfavorable medical occurrence, including any abnormal physical exam or laboratory finding, symptom, or disease, temporally associated with the participant's participation in the research. Patients were queried for hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions.
Groups:
- 12 SSc Participants Placebo: 12 SSc participants were studied 5 hours after oral placebo administration (10 mg/kg body mass)
- 12 SSc Participants BH4: 12 SSc participants were studied 5 hours after oral BH4 administration (10 mg/kg body mass)
Arm/Group | 12 SSc Participants Placebo | 12 SSc Participants BH4
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
This trial was initially intended to include 32 patients with SSc with and without clinical complications of SSc randomly assigned oral BH4 or placebo for 5 consecutive days in a double-blind randomized crossover design. Due to budget constraints, we adapted the design to studying 12 patients, 5 hours after oral BH4 administration (10 mg/kg body weight) or placebo on separate days using controlled, counterbalanced, double-blind, crossover experimental design and a five day wash-out period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (5):
  • Study Protocol: 38705 SSc Registry Trial (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT02530996/Prot_000.pdf
  • Study Protocol: 40212 (12 patients) (2015-03-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT02530996/Prot_001.pdf
  • Statistical Analysis Plan (2016-04-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT02530996/SAP_002.pdf
  • Informed Consent Form: 38705 (156 patients) (2020-08-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT02530996/ICF_003.pdf
  • Informed Consent Form: 40212 (12 patients) (2015-05-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT02530996/ICF_004.pdf